CLINICAL TRIAL: NCT02659072
Title: Infectious Risk of Vaginal Ultrasound Examination: Evaluation and Modeling From Human Papillomavirus (HPV)
Acronym: PREEV
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI14013
Record Dates: First submitted 2016-01-05; First posted 2016-01-20 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: GYNAECOLOGICAL INFECTION

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multicenter observational survey of the presence of Human Papilloma Virus (HPV) on trans vaginal ultrasound (TVUS) probes, and of the behavior of professionals during US examination and probe disinfection. This will allow modeling the risk of HPV transmission, and could contribute establishing future guidelines for reducing the risk of transmission of microorganisms and the risk of infection through TVS.

DETAILED DESCRIPTION:
Prevention of infection Endo Vaginal sonography. Brief Summary

Background Trans vaginal sonography (TVS) is widely used in obstetrics and gynecology. Because of the relative lack of data, there is no universal agreement on how to prevent the transmission of pathogens and the risk of infection through TVS. Whereas American guideline are more stringent, French health authorities recommend low-level disinfection of the probe between two patients with the use of probe cover, and intermediate level disinfection at least once daily and in case of visible contamination of the probe, or rupture of the probe cover. For the coupling gel, guidelines do not agree on whether or not it should be sterile.

Transmitting infectious agents may result from a variety of causes: failure to disinfect the probe, contaminated gel, contamination of the probe cover due to incorrect manipulation and failure to comply with hand washing or disinfection.

Due to resistance to disinfection, high prevalence, and potential oncogenic role, we will use HPV as a marker for the presence of pathogens on the probe, the probe cover, and the environment.

Objectives Primary objective: to assess the presence of HPV on bare probes and on probes with their probe-cover in routine practice

Secondary objectives:

1. - To assess compliance to guidelines of prevention of pathogens
2. - To identify factors associated with the presence of HPV on the probe

2a Factors related to the procedure Compliance to disinfection guidelines prior to performing TVS Rank of procedure since last daily midlevel disinfection Presence of HPV on the ultrasound machine key board, a proxy of the environment 2b Factors related to the center in which TVS is performed Compliance to daily disinfection guidelines Traceability of the disinfection processes Type of center (emergency clinic /planned sessions / obstetrics / gynecology /IVF monitoring) 3 - To estimate the incidence of probe cover rupture and of visible probe contamination by bodily fluids 4 - To model the cost effectiveness of strategies of disinfection

Methods Type of study: observational survey

Main outcome criterion:

Percentage and 95 % confidence interval of TVS procedure

* with bare probe positive for HPV
* with covered probe positive for HPV Statistical unit: each procedure surveyed Viral assays HPV DNA detection will be performed on all samples (keyboard, bare and covered probe) using the cobas® HPV Test Kit (Roche): This test allows to detect the presence of cellular DNA and DNA of 14 high-risk HPV (genotypes 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68) and to specifically identify the presence of HPV16 and 18. In case of positive result for both bare and covered probe, a detection of HPV complete episomal genome will be performed, and circular HPV DNA will be amplified using a polymerase whch selectively amplifies circular double-stranded DNA with specific degenerate HPV primers. The amplicons will then be sequenced using specific HPV primers GP5 + / GP6 + (MARINCEVIC Y-Zuniga et al, 2012, Virology).

Secondary outcome criteria Percentage of procedures with keyboard positive for HPV Percentage of procedures with visible rupture of probe cover Percentage of procedures with visibly tainted probes Percentage of procedures with visible rupture of probe cover during previous procedure Percentage of procedures with visibly tainted probes during previous procedure Percentage of presence of each disinfection guideline item since last procedure and before the probe is tested for the presence of HPV Percentage of centers with a written protocol complying with disinfection guidelines Percentage of centers with traceability of disinfection procedures.

Number of observations: 1000 TVS procedures

Inclusion criterion: Any TVS performed in a participating center during an observation session Exclusion criteria: TVS with invasive procedure. Patient refusal Center selection: private and public centers from the Ile de France region, performing TVS routinely, who volunteered to enroll.

Perspectives Evaluating the presence of HPV on TVS probes in relation with the actual behavior of professionals in routine practice will help us modeling the risk of transmitting pathogens during TVS and may contribute to establishing prevention guidelines

ELIGIBILITY:
Inclusion Criteria:

* All examination of endo-vaginal ultrasound performed at participating center during a predetermined observation session,

Exclusion Criteria:

* * Endo-Vaginal ultrasound with invasive procedure (with cutaneous or mucosal break)

  * Refusal of the patient that non-personal data are addressed in a study,

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women who will have an examination of endo-vaginal ultrasound
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Percentage and 95 % confidence interval of TVS procedures with bare probe positive for HPV | 12 months
  Qualitative variable. Statistical unit: each procedure surveyed
Percentage and 95 % confidence interval of TVS procedures with covered probe positive for HPV | 12 months
  Qualitative variable. Statistical unit: each procedure surveyed

SECONDARY OUTCOMES:
Percentage of procedures with keyboard positive for HPV | 12 months
  Qualitative variables will be analyzed as percentages of presence. Statistical unit: each procedure surveyed. In addition, the number of disinfection items present will be added as a score.
Percentage of procedures with visible rupture of probe cover | 12 months
  Qualitative variables will be analyzed as percentages of presence. Statistical unit: each procedure surveyed. In addition, the number of disinfection items present will be added as a score.
Percentage of procedures with visibly tainted probes | 12 months
  Qualitative variables will be analyzed as percentages of presence. Statistical unit:
Percentage of procedures with visible rupture of probe cover during previous procedure | 12 months
  Qualitative variables will be analyzed as percentages of presence. Statistical unit:
Percentage of procedures with visibly tainted probes during previous procedure | 12 months
  Qualitative variables will be analyzed as percentages of presence. Statistical unit:
Percentage of presence of each disinfection guideline item since last procedure and before the probe is tested for the presence of HPV | 12 months
  Qualitative variables will be analyzed as percentages of presence. Statistical unit:
Percentage of centers with a written protocol complying with disinfection guidelines | 12 months
  Qualitative variables will be analyzed as percentages of presence. Statistical unit:
percentage of centers with traceability of disinfection procedures. | 12 months
  Qualitative variables will be analyzed as percentages of presence. Statistical unit:

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe LUCET, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital La Pitié Salpêtrire, Paris, France